CLINICAL TRIAL: NCT01833143
Title: A Phase 2 Trial of Bortezomib in KRAS-Mutant Non-Small Cell Lung Cancer in Never Smokers or Those With KRAS G12D
Brief Title: Bortezomib in KRAS-Mutant Non-Small Cell Lung Cancer in Never Smokers or Those With KRAS G12D
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-222
Record Dates: First submitted 2013-04-11; First posted 2013-04-16 (Estimated); Results first posted 2020-07-23 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2019-08

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: KRAS-Mutant; Bortezomib; KRAS G12D; 12-222
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bortezomib; Acyclovir

ARMS (1):
- Bortezomib (Experimental): Bortezomib will be administered by subcutaneous injection twice weekly for 2 weeks (Days 1, 4, 8, and 11) at 1.3 mg/m2/dose followed by a 10-day rest period for a 21 day cycle. Dose modifications are permitted as per a prescribed algorithm. Acyclovir at 400mg daily is recommended as prophylaxis for herpes zoster. Restaging scans, with evaluation of response, will be done every 2 cycles (6 weeks of treatment ± 7 days). Treatment will continue until clinical disease progression, unacceptable toxicity, treatment delay > 2 weeks, or at the discretion of the treating physician or patient.
  Interventions: Drug: Bortezomib; Drug: Acyclovir

INTERVENTIONS:
Drug: Bortezomib
Drug: Acyclovir

SUMMARY:
The purpose of this study is to test the drug Bortezomib to see how well it works. The investigators want to find out what effects, good or bad, it has on patients with a limited smoking history or who have a specific mutation associated with their lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic or cytologic evidence of non-small cell lung cancer (NSCLC)
* Documented KRAS mutation
* History of smoking < 100 cigarettes (never-smoker) OR patient with a KRAS G12D mutation regardless of smoking history
* Clinical stage IIIB/IV or recurrent/medically inoperable NSCLC
* Age ≥ 18 years
* Three (3) weeks since last chemotherapy, and three (3) weeks since prior radiation therapy and recovered from treatment
* Karnofsky performance status ≥ 70%
* Adequate hematologic, and/or hepatic function WBC ≥ 3,000/ul or absolute neutrophil count ≥ 1,000/ul Hemoglobin ≥ 9.0 g/dl Platelet count ≥ 100,000/ul AST ≤ 2.0 X ULN (upper limit of normal)
* Total bilirubin ≤1.5 x ULN Measurable indicator lesions by RECIST v1.1 criteria.
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Female subject is either postmenopausal for at least 1 year before the screening visit, is surgically sterilized or if they are of childbearing potential, agree to practice 2 effective methods of contraception from the time of signing the informed consent form through 30 days after the last dose of bortezomib, or agree to completely abstain from heterosexual intercourse.
* Male subjects must agree to 1 of the following: practice effective barrier contraception during the entire study treatment period and through a minimum of 30 days after the last dose of study drug, or completely abstain from heterosexual intercourse.

Exclusion Criteria:

* Uncontrolled central nervous system metastases defined as any lesion which is either a. symptomatic, or requiring escalating doses of corticosteroids
* Significant medical history or unstable medical condition such as uncontrolled diabetes myocardial infarction within 6 months prior to enrollment New York Heart Association Class III or IV heart failure severe uncontrolled ventricular arrythmias uncontrolled angina ECG evidence of acute ischemia or active conduction system abnormalities
* Baseline ≥ grade 2 peripheral neuropathy by CTCAE v 4.0 (Appendix B)
* Known hypersensitivity to boron or mannitol
* Female patients who are pregnant/lactating or have a positive serum or urine β-hCG pregnancy test
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* No active concurrent malignancy, with the exception of in-situ malignancy completely resected basal cell carcinoma or squamous cell carcinomas of the skin low-risk prostate cancer after curative therapy
* Participation in clinical trials with other investigational agents not included in this trial, within 14 days of the start of this trial and throughout the duration of this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-04-11 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Riely, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center at Phelps, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bortezomib
Started | 17
Completed | 16
Not Completed | 1
Not completed — Not Treated | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bortezomib
Number analyzed (Participants) | 17
Age, Continuous [Median (Full Range); unit: years] | 67 [36 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 13
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Response Rate
Description: The following evaluations will be conducted to assess the efficacy of bortezomib - radiographic response rate by RECIST v1.1. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Bortezomib
Number analyzed (Participants) | 17
Participants
  Partial Response | 1
  Stable Disease | 6
  Progression of Disease | 10

2. Secondary Outcome: Progression Free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bortezomib
Number analyzed (Participants) | 17
months | 1 [1 to 6]

3. Secondary Outcome: Participants Evaluated for Toxicity
Description: Before each drug dose, the patient will be evaluated for possible toxicities that may have occurred after the previous dose(s). Toxicities are to be assessed according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE v4.0,).
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Bortezomib
Number analyzed (Participants) | 17
Participants | 17

4. Secondary Outcome: Overall Survival
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bortezomib
Number analyzed (Participants) | 17
months | 13 [6 to 30]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Bortezomib
All-Cause Mortality (participants affected / at risk) | 12/17
Serious Adverse Events (participants affected / at risk) | 4/17
Other Adverse Events (participants affected / at risk) | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib (N=17)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Fever (General disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib (N=17)
Fatigue (General disorders) | 8
Diarrhea (Gastrointestinal disorders) | 6
Anorexia (Metabolism and nutrition disorders) | 4
Constipation (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 4
Papulopustular rash (Skin and subcutaneous tissue disorders) | 4
Headache (Nervous system disorders) | 3
Localized edema (General disorders) | 3
Fever (General disorders) | 2
Injection site reaction (General disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 2
Peripheral motor neuropathy (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2
Platelet count decreased (Investigations) | 2
Vomiting (Gastrointestinal disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Depression (Psychiatric disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Eye pain (Eye disorders) | 1
Flu like symptoms (General disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-02-07): https://cdn.clinicaltrials.gov/large-docs/43/NCT01833143/Prot_SAP_000.pdf